CLINICAL TRIAL: NCT01492400
Title: Safety and Efficacy Study of Dexamethasone Versus Ranibizumab in Patients With Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 206207-024
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Results first posted 2015-01-29 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Dexamethasone; Calcium Dobesilate; Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexamethasone Intravitreal Implant (Experimental): Injection of 700 ug dexamethasone intravitreal implant into the study eye on Day 1, Month 5, and Month 10.
  Interventions: Drug: dexamethasone Intravitreal Implant
- ranibizumab (Active Comparator): Injection of ranibizumab 0.5 mg into the study eye on Day 1. Patients may receive additional injections on a monthly basis, as needed, for disease progression.
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: dexamethasone Intravitreal Implant — Injection of 700 ug dexamethasone intravitreal implant into the study eye on Day 1, Month 5, and Month 10.
  Other Names: Ozurdex®
  Arms: dexamethasone Intravitreal Implant
Drug: ranibizumab — Injection of ranibizumab 0.5 mg into the study eye on Day 1. Patients may receive additional injections on a monthly basis, as needed, for disease progression.
  Other Names: Lucentis®
  Arms: ranibizumab

SUMMARY:
This study will compare the safety and efficacy of the 700 ug dexamethasone intravitreal implant with ranibizumab 0.5 mg intravitreal injections in patients with diabetic macular edema (DME).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 or 2 diabetes mellitus
* Diagnosis of macular edema
* Visual acuity between 20/200 to 20/40

Exclusion Criteria:

* Eye surgery to the study eye within 3 months
* Use of Ozurdex® within 9 months
* Any active ocular inflammation and infection
* Diagnosis of glaucoma
* Use of anti-VEGF treatment (e.g., Lucentis®) within 3 months in the eye or systemic use (e.g., Avastin®) within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2012-03-09 (Actual); Primary Completion 2014-02-13 (Actual); Study Completion 2014-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (13):
- Arlington, Texas, United States
- Brussels, Belgium
- Denmark (2):
  - Copenhagen
  - Glostrup Municipality
- Paris, France
- Ahaus, Germany
- Tel Aviv, Israel
- Udine, Italy
- Nijmegen, Netherlands
- Coimbra, Portugal
- Pretoria, South Africa
- Barcelona, Spain
- London, England, United Kingdom

REFERENCES:
- [Background] Callanan DG, Loewenstein A, Patel SS, Massin P, Corcostegui B, Li XY, Jiao J, Hashad Y, Whitcup SM. A multicenter, 12-month randomized study comparing dexamethasone intravitreal implant with ranibizumab in patients with diabetic macular edema. Graefes Arch Clin Exp Ophthalmol. 2017 Mar;255(3):463-473. doi: 10.1007/s00417-016-3472-1. Epub 2016 Sep 8. PMID 27632215
- [Derived] Rittiphairoj T, Mir TA, Li T, Virgili G. Intravitreal steroids for macular edema in diabetes. Cochrane Database Syst Rev. 2020 Nov 17;11(11):CD005656. doi: 10.1002/14651858.CD005656.pub3. PMID 33206392
- [Derived] Chakravarthy H, Devanathan V. Molecular Mechanisms Mediating Diabetic Retinal Neurodegeneration: Potential Research Avenues and Therapeutic Targets. J Mol Neurosci. 2018 Nov;66(3):445-461. doi: 10.1007/s12031-018-1188-x. Epub 2018 Oct 6. PMID 30293228

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone Intravitreal Implant | Ranibizumab
Started | 181 | 182
Completed | 165 | 166
Not Completed | 16 | 16
Not completed — Miscellaneous Reasons | 2 | 3
Not completed — Personal Reasons | 0 | 5
Not completed — Lost to Follow-up | 3 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Adverse Event | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone Intravitreal Implant | Ranibizumab | Total
Number analyzed (Participants) | 181 | 182 | 363
Age, Customized [Number; unit: Participants]
  <45 years | 5 | 5 | 10
  45 to 65 years | 102 | 96 | 198
  >65 years | 74 | 81 | 155
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 66 | 135
  Male | 112 | 116 | 228

OUTCOME MEASURES:

1. Primary Outcome: Average Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The average BCVA is calculated across study visits for each patient. A positive number change from baseline indicates an improvement and a negative number change from baseline indicates a worsening.
Time Frame: Baseline, 12 Months
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Dexamethasone Intravitreal Implant | Ranibizumab
Number analyzed (Participants) | 181 | 182
Letters
  Baseline | 60.2 (9.74) | 60.4 (9.34)
  Change from Baseline at 12 Months | 4.34 (7.342) | 7.60 (6.735)

2. Secondary Outcome: Change From Baseline in Foveal Thickness Measured by Optical Coherence Tomography (OCT) in the Study Eye
Description: OCT is a laser based non-invasive diagnostic system providing high-resolution imaging sections of the fovea (part of the retina) in the study eye after pupil dilation. A negative change from baseline indicates an improvement (less foveal thickness) and a positive change from baseline indicates a worsening (more foveal thickness).
Time Frame: Baseline, Month 12
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Dexamethasone Intravitreal Implant | Ranibizumab
Number analyzed (Participants) | 181 | 182
Microns
  Baseline | 465.1 (136.09) | 471.2 (139.51)
  Change from Baseline at Month 12 (N=163, 166) | -173.9 (129.64) | -163.5 (161.34)

3. Secondary Outcome: Change From Baseline in Total Area of Macular Leakage in the Study Eye Measured on Fluorescein Angiography (FA)
Description: FA is a technique for examining the circulation of the retina (and detecting any leakage) using a dye-tracing method. Photographs are taken with a specialized low-power microscope with an attached camera designed to photograph the interior of the eye, including the retina and optic disc. A negative change from baseline indicates a decrease in leakage (improvement) and a positive change from baseline indicates an increase in leakage (worsening).
Time Frame: Baseline, Month 12
Population: Intent-to-Treat: all randomized patients
Measure: Mean (Standard Deviation); unit: Square Millimeters (mm^2)
Arm/Group | Dexamethasone Intravitreal Implant | Ranibizumab
Number analyzed (Participants) | 172 | 177
Square Millimeters (mm^2)
  Baseline | 19.2 (13.01) | 18.9 (12.55)
  Change from Baseline at Month 12 (N=125, 142) | -16.1 (11.64) | -12.0 (10.54)

ADVERSE EVENTS:
Description: Treatment emergent adverse events (TEAE) are reported and include all adverse events (AEs) and serious adverse events (SAEs) that began or worsened after study treatment.
Arm/Group | Dexamethasone Intravitreal Implant | Ranibizumab
Serious Adverse Events (participants affected / at risk) | 40/181 | 41/182
Other Adverse Events (participants affected / at risk) | 160/181 | 104/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Dexamethasone Intravitreal Implant (N=181) | Ranibizumab (N=182)
Renal Failure Acute (Renal and urinary disorders) | 4 | 3
Cardiac Failure Congestive (Cardiac disorders) | 4 | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Coronary Artery Disease (Cardiac disorders) | 2 | 2
Sepsis (Infections and infestations) | 2 | 2
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1
Chest Pain (General disorders) | 2 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 2 | 0
Intraocular Pressure Increased (Investigations) | 2 | 0
Syncope (Nervous system disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Angina Pectoris (Cardiac disorders) | 1 | 2
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Cardiac Failure (Cardiac disorders) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 1
Diabetic Foot (Skin and subcutaneous tissue disorders) | 1 | 1
Endophthalmitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Renal Failure Chronic (Renal and urinary disorders) | 1 | 1
Wound Infection (Infections and infestations) | 1 | 1
Abscess Limb (Infections and infestations) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0
Anal Abscess (Infections and infestations) | 1 | 0
Asthenia (General disorders) | 1 | 0
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac Pacemaker Insertion (Surgical and medical procedures) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Grand Mal Convulsion (Nervous system disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Kidney Infection (Infections and infestations) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Liposuction (Surgical and medical procedures) | 1 | 0
Local Swelling (General disorders) | 1 | 0
Lung Squamous Cell Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mantle Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningorrhagia (Nervous system disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Open Angle Glaucoma (Eye disorders) | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/112 | 0/116
Pyelonephritis (Infections and infestations) | 1 | 0
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Sialoadenitis (Infections and infestations) | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Squamous Cell Carcinoma of the Tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 2
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 2
Myocardial Ischaemia (Cardiac disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 2
Abdominal Wall Abscess (Infections and infestations) | 0 | 1
Aortic Valve Stenosis (Cardiac disorders) | 0 | 1
Atypical Pneumonia (Infections and infestations) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Choroiditis (Eye disorders) | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0/69 | 1/66
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 1
Generalised Oedema (General disorders) | 0 | 1
Haemorrhagic Stroke (Nervous system disorders) | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypertensive Crisis (Vascular disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Infected Bites (Infections and infestations) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Lacrimation Increased (Eye disorders) | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Nephropathy (Renal and urinary disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 0 | 1
Peripheral Vascular Disorder (Vascular disorders) | 0 | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Septic Shock (Infections and infestations) | 0 | 1
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sudden Hearing Loss (Ear and labyrinth disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Ventricular Tachyarrhythmia (Cardiac disorders) | 0 | 1
Vitreous Haemorrhage (Eye disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Weight Decreased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexamethasone Intravitreal Implant (N=181) | Ranibizumab (N=182)
Anaemia (Blood and lymphatic system disorders) | 6 | 10
Conjunctival Haemorrhage (Eye disorders) | 36 | 24
Cataract (Eye disorders) | 28 | 8
Vitreous Haemorrhage (Eye disorders) | 22 | 7
Visual Acuity Reduced (Eye disorders) | 14 | 5
Cataract Subcapsular (Eye disorders) | 14 | 1
Vitreous Floaters (Eye disorders) | 13 | 2
Ocular Hypertension (Eye disorders) | 11 | 2
Eye Pain (Eye disorders) | 10 | 6
Diabetic Retinal Oedema (Eye disorders) | 10 | 5
Vitreous Detachment (Eye disorders) | 10 | 5
Punctate Keratitis (Eye disorders) | 9 | 3
Macular Oedema (Eye disorders) | 3 | 10
Influenza (Infections and infestations) | 9 | 4
Intraocular Pressure Increased (Investigations) | 65 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.